CLINICAL TRIAL: NCT02477176
Title: A Prospective, Multicenter Study Investigating Reherniation Risk Factors and Associated Costs in Primary Lumbar Disc Herniation Patients
Brief Title: Lumbar Discectomy Control Study, Risk Factors for Reherniation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: US CONTROL-001
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Spine Disc Herniation
MeSH Terms: interventions — Diskectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Small annular defect group: Patients with lumbar defect less than 6mm wide after lumbar discectomy
  Interventions: Other: Discectomy
- Large annular defect group: Patients with lumbar defect greater than 6mm wide after lumbar discectomy
  Interventions: Other: Discectomy

INTERVENTIONS:
Other: Discectomy — Lumbar discectomy

SUMMARY:
The purpose of this 12-month, prospective, multicenter study is to investigate the effect of annular defect size and other risk factors on reherniation and associated costs in primary lumbar discectomy patients.

DETAILED DESCRIPTION:
This study will enroll up to 100 patients at select US (approximately 4-7) sites. Patients that are scheduled for an L1-S1 discectomy and who meet the pre-operative eligibility criteria will be considered for study participation. Patients will be divided into two arms (small- and large-defect) based on the size of their annular defect as measured intra-operatively; each arm will be capped at 50 patients. All patients included in the trial will be followed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 75 years old and skeletally mature (male or female).
2. Patients with posterior or posterolateral disc herniations at one level between L1 and S1 with radiographic confirmation of neural compression using MRI. [Note: Intraoperatively, only patients with an annular defect (post discectomy) between 4mm and 6mm tall and 6mm and 10mm wide shall qualify.]
3. Radiculopathy (with or without back pain) with a positive Straight Leg Raise (0 - 60 degrees)22 (L45, L5S1) or Femoral Stretch Test (L12, L23, L34)
4. Oswestry Questionnaire score of at least 40/100 at baseline.
5. VAS leg pain (one or both legs) of at least 40/100 at baseline.
6. Psychosocially, mentally and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.
7. Minimum posterior disc height of 5mm at the index level.

Exclusion Criteria:

1. Spondylolisthesis Grade II or higher (25% slip or greater).
2. Subject requires spinal surgery other than a discectomy (with or without laminotomy) to treat leg/back pain (scar tissue and osteophyte removal is allowed).
3. Subject has back or non-radicular leg pain of unknown etiology.
4. Prior surgery at the index lumbar vertebral level.
5. Subject requiring a spine dual energy x-ray absorptiometry (i.e., patients with SCORE of ≥ 6) with a T Score less than -2.0 at the index level. For patients with a herniation at L5/S1, the average T score of L1-L4 shall be used.
6. Subject has clinically compromised vertebral bodies in the lumbosacral region due to any traumatic, neoplastic, metabolic, or infectious pathology.
7. Subject has sustained pathologic fractures of the vertebra or multiple fractures of the vertebra or hip.
8. Subject has scoliosis of greater than ten (10) degrees (both angular and rotational).
9. Any metabolic bone disease.
10. Subject has an active infection either systemic or local.
11. Subject has cauda equine syndrome or neurogenic bowel/bladder dysfunction.
12. Subject has severe arterial insufficiency of the legs or other peripheral vascular disease. (Screening on physical examination for patients with diminution or absence of dorsalis pedis or posterior tibialis pulses. If diminished or absent by palpation, then an arterial ultrasound is required with vascular plethysmography. If the absolute arterial pressure is below 50mm of Hg at the calf or ankle level, then the patient is to be excluded.)
13. Subject has significant peripheral neuropathy, patient defined as a patient with Type I or Type II diabetes or similar systemic metabolic condition causing decreased sensation in a stocking-like or non-radicular and non-dermatomal distribution in the lower extremities.
14. Subject has insulin-dependent diabetes mellitus.
15. Subject is morbidly obese (defined as a body mass index >40, or weighs more than 100 lbs over ideal body weight).
16. Subject has been diagnosed with active hepatitis, AIDS, or HIV.
17. Subject has been diagnosed with rheumatoid arthritis or other autoimmune disease.
18. Subject has active tuberculosis or has had tuberculosis in the past three (3) years.
19. Subject has a history of active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no signs or symptoms of the malignancy for at least two (2) years.
20. Subject is immunologically suppressed, received steroids >1 month over the past year.
21. Currently taking anticoagulants, other than aspirin, unless the patient can be taken off the anticoagulant for surgery.
22. Subject has a current chemical/alcohol dependency or significant psychosocial disturbance.
23. Subject has a life expectancy of less than three (3) years.
24. Subject is currently involved in active spinal litigation.
25. Subject is currently involved in another investigational study.
26. Subject is incarcerated.
27. Patients will be divided into two arms (small- and large-defect) based on the width of their annular defect as measured intra-operatively. Patients with defects <6mm in width will be in the "small defect" arm; patients with defects ≥6mm in width will be in the "large defect" arm. Each arm will be capped at 50 patients. Once 50 patients are accrued in one arm, subsequent patients who meet the criteria for that arm will be excluded. Enrollment will continue until both arms are filled.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with single level, symptomatic lumbar disc herniation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02-17 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Lumbar reherniation at the index level | 12 Months
  Reherniation of index level, yes or no

SECONDARY OUTCOMES:
Reoperation at the index level | 12 Months
  Reoperation at index level, yes or no
Hospitalization at physician cost | 12 Months
  The total hospitalization and physician costs for the index surgery and any secondary surgical intervention of the index level will be summed and reported for each subject based on data collected on the UB-04

CONTACTS AND LOCATIONS:
Overall Officials: David H Kim, MD, Study Chair — New England Baptist Hospital
Locations (4):
- United States (4):
  - Midwest Orthopaedics at Rush Medical Center, Chicago, Illinois
  - Orthopaedic Specialists Of The Four States, Galena, Kansas
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Michigan Orthopedic Specialists, Dearborn, Michigan